CLINICAL TRIAL: NCT07215039
Title: Improving Prison Health Equity Through Cancer Literacy and Screening Awareness in Florida
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Radiation Oncology Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: MC250903; NCI-2025-05529 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25-003194 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2025-10-08; First posted 2025-10-10 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Participants complete a survey on study.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Non-interventional study

SUMMARY:
This study evaluates cancer screening awareness, personal and family cancer history, and barriers to screening among incarcerated women at Gadsden Correctional Facility. The information will be used to inform the content of a tailored digital educational module on screenable types of cancer, their risk factors, and current screening guidelines that will be disseminated to US prisons and incorporated into release programs and general health literacy programs.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18+ currently incarcerated at Gadsden Correctional Facility
* Pregnant participants are allowed

Exclusion Criteria:

* Women under 18 or not incarcerated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women currently incarcerated at Gadsden Correctional Facility
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Self-reported cancer screening history | Baseline (completion of survey)
  Assessed as the proportion of incarcerated women who meet national cancer screening guidelines based on self-reported screening history. Participants will complete a 4-page, paper-based, anonymous survey that should take approximately 15 minutes to complete. The survey consists of mainly yes/no questions with a few multiple choice and open-ended questions. This is a qualitative survey used to record basic demographic information, cancer knowledge, risk factors, screening history, and adherence to preventive cancer care. Survey results will be used to inform the content of a tailored digital educational module on screenable types of cancer, their risk factors, and current screening guidelines.

SECONDARY OUTCOMES:
Awareness of cancer risk factors | Baseline (completion of survey)
  Participants will complete a 4-page, paper-based, anonymous survey that should take approximately 15 minutes to complete. The survey consists of mainly yes/no questions with a few multiple choice and open-ended questions. This is a qualitative survey used to record basic demographic information, cancer knowledge, risk factors, screening history, and adherence to preventive cancer care. Survey results will be used to inform the content of a tailored digital educational module on screenable types of cancer, their risk factors, and current screening guidelines.
Awareness of cancer screening guidelines | Baseline (completion of survey)
  Participants will complete a 4-page, paper-based, anonymous survey that should take approximately 15 minutes to complete. The survey consists of mainly yes/no questions with a few multiple choice and open-ended questions. This is a qualitative survey used to record basic demographic information, cancer knowledge, risk factors, screening history, and adherence to preventive cancer care. Survey results will be used to inform the content of a tailored digital educational module on screenable types of cancer, their risk factors, and current screening guidelines.
Barriers to cancer screening within correctional settings | Baseline (completion of survey)
  Participants will complete a 4-page, paper-based, anonymous survey that should take approximately 15 minutes to complete. The survey consists of mainly yes/no questions with a few multiple choice and open-ended questions. This is a qualitative survey used to record basic demographic information, cancer knowledge, risk factors, screening history, and adherence to preventive cancer care. Survey results will be used to inform the content of a tailored digital educational module on screenable types of cancer, their risk factors, and current screening guidelines.
Barriers to cancer screening follow-up within correctional settings | Baseline (completion of survey)
  Participants will complete a 4-page, paper-based, anonymous survey that should take approximately 15 minutes to complete. The survey consists of mainly yes/no questions with a few multiple choice and open-ended questions. This is a qualitative survey used to record basic demographic information, cancer knowledge, risk factors, screening history, and adherence to preventive cancer care. Survey results will be used to inform the content of a tailored digital educational module on screenable types of cancer, their risk factors, and current screening guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Oluwadamilola T. Oladeru, MD, MBA, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials